CLINICAL TRIAL: NCT00357136
Title: Online Survey on Computer Password Usage.
Status: Completed | Type: Observational
Sponsor: Towson University (Other)
Responsible Party: Sponsor
Other Study IDs: 888
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Behavioral: password usage

SUMMARY:
Researchers at Towson University are conducting a study of computer password behaviors among users who have difficulty using their hands and arms (e.g., individuals with carpal tunnel syndrome, high level spinal cord injuries, etc.). Volunteers are needed to take a short 5-10 minute online survey.

The survey is completely confidential and anonymous. If you would like to participate, please visit the URL below. Thank you.

http://pages.towson.edu/jdarcy/securitysurvey.htm

DETAILED DESCRIPTION:
Two researchers from the Department of Computer & Information Sciences at Towson University are seeking individuals who have difficulty using their hands and arms (e.g., as result of carpal tunnel syndrome, high level spinal cord injuries, etc.) to participate in a survey. The survey should take approximately 10 minutes to complete and all responses will remain completely confidential and anonymous.

The purpose of the survey is to gain insight into the computing behaviors of individuals with upper-body motor impairments. We expect that the results will help researchers and system developers create more effective access control techniques to meet the special needs of this user population. The results should also assist employers in providing improved technical and procedural support to computer users that have difficulties using standard input devices.

If you would like to take the online survey, please go to the following link:

http://www.towson.edu/cosc/securitysurvey

If you prefer a paper version of the survey, please send us an e-mail that contains your mailing address and we will send the survey to you.

Contact information:

John D'Arcy, Ph.D. (jdarcy@towson.edu) Jinjuan Feng, Ph.D. (jfeng@towson.edu) Department of Computer & Information Sciences Towson University 7800 York Road Towson, MD 21252 U.S.A.

ELIGIBILITY:
Inclusion Criteria:

* Users who have difficulty using their hands or arms

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-07; Primary Completion 2006-12 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinjuan Feng, Ph. D., Principal Investigator — Towson University
Locations (1):
- Towson University, Towson, Maryland, United States